CLINICAL TRIAL: NCT03516604
Title: The Effects of PF-04995274 on Emotional Processing in Un-medicated Depressed Patients
Brief Title: PF-04995274 and Emotional Processing in Un-medicated Depression
Acronym: RESTAND
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council (Other Government); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PF04995274 Study 1 RESTAND; MR/P012604/1 (Other Grant/Funding Number: MRC (UK))
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Depression, Unipolar
MeSH Terms: conditions — Depressive Disorder | interventions — Citalopram; Dexetimide

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of three groups (PF-04995264, citalopram or placebo) and receive their allocated study medication for 7 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PF-04995274 (Experimental): PF-04995274, three x 5mg tablet (15mg total), once daily for 7-9 days
  + 1 placebo capsule, once daily for 7-9 days
  Interventions: Drug: PF-04995274; Drug: Placebo oral capsule
- Citalopram (Active Comparator): Citalopram, one x 20mg capsule, once daily for 7-9 days
  + 3 placebo tablets, once daily for 7-9 days
  Interventions: Drug: Citalopram; Drug: Placebo Oral Tablet
- Placebo (Placebo Comparator): 3 placebo tablets and 1 placebo capsule, once daily for 7-9 days
  Interventions: Drug: Placebo Oral Tablet; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: PF-04995274 — PF-04995274 tablets
  Arms: PF-04995274
Drug: Citalopram — Citalopram capsule
  Other Names: Celexa, Cipramil
  Arms: Citalopram
Drug: Placebo Oral Tablet — Placebo tablet, identical to PF-04995274 tablet
  Arms: Citalopram; Placebo
Drug: Placebo oral capsule — Placebo capsule, identical to citalopram capsule
  Arms: PF-04995274; Placebo

SUMMARY:
This study will test whether seven days administration of a serotonin receptor subtype 4 (5HT4) agonist called PF-04995274 has positive effects on cognition, emotional processing and neural activity in unmedicated depressed patients compared to placebo. The study will also include a group of patients randomised to seven days administration of citalopram (20 mg), which is a standard treatment for depression.

DETAILED DESCRIPTION:
This study uses a double-blind, placebo-controlled, randomised between-groups design to test if administration of a serotonin receptor subtype 4 (5HT4) agonist called PF-04995274 has positive effects on emotional processing and neural activity in unmedicated depressed patients. Participants are patients who fulfill criteria for current episode of Major Depressive Disorder (MDD), and they will be randomised to receive 7 days treatment with either PF-04995274 (15 mg daily), citalopram (20 mg daily) or a matched placebo. Participants will come for a Screening Visit, a First Dose Visit, Research Visit One (including MRI scan) and Research Visit Two (including measures of emotional processing and non-emotion cognition).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-65 years;
* Willing and able to give informed consent for participation in the study;
* Sufficiently fluent English to understand and complete the tasks;
* Registered with a GP and consents to GP being informed of participation in study;
* Meet DSM-V criteria for current Major Depressive Disorder [as determined by the Structured Clinical interview for DSM-V (SCID)];
* Participant must have received no drug or face-to-face psychological treatment for the current episode of depression/ in the previous six weeks;
* Participants engaging in sex with a risk of pregnancy must agree to use a highly effective method of contraception from Screening Visit until 30 days after receiving study medication treatment, female participants must not breastfeed, and male participants must not donate sperm.

Exclusion Criteria:

* History of or current DSM-V bipolar disorder, schizophrenia or eating disorders. Participants who fulfil current criteria for other comorbid disorders may still be entered into the study, if, in the opinion of the Investigator, the psychiatric diagnosis will not compromise safety or affect data quality;
* First-degree relative with a diagnosis of Bipolar Disorder type 1;
* Current usage of psychotropic medication;
* Failure to respond to antidepressant medication in current episode;
* Electroconvulsive therapy for the treatment of the current episode of depression;
* Participants undergoing any form of face-to-face structured psychological treatment during the study;
* Clinically significant abnormal values for liver function tests, clinical chemistry, urine drug screen, blood pressure measurement and ECG. A participant with a clinical abnormality or parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures;
* History of stimulant abuse (lifetime; e.g. amphetamine, cocaine), or of alcohol abuse within one year or of alcohol dependence within the lifetime;
* History of, or current medical conditions which in the opinion of the investigator may interfere with the safety of the participant or the scientific integrity of the study, including epilepsy/seizures, brain injury, severe hepatic or renal disease, severe gastro-intestinal problems, Central Nervous System (CNS) tumors, severe neurological problems (like Parkinson's; blackouts requiring hospitalisation);
* Medical conditions that may alter the hemodynamic parameters underlying the BOLD signal (e.g., inadequately treated hypertension, diabetes mellitus);
* Clinically significant risk of suicide;
* Current pregnancy (as determined by urine pregnancy test taken during Screening and First Dose Visits), breastfeeding or planning a pregnancy during the course of the study;
* Participant not willing to use a suitable method of contraception for 30 days after receiving study drug treatment;
* Any contraindication to MRI scanning (e.g. metal objects in body, pacemakers, significant claustrophobia, pregnancy);
* Participants with Body Mass Index (BMI) outside the 18 to 36 kg/m2 range at the Screening Visit.
* Night-shift working or recent travel involving significant change of timezones;
* Excessive caffeine consumption, i.e., consumption higher than 8 cups of standard caffeinated drinks (tea, instant coffee) or higher than 6 cups of stronger coffee or other drinks containing methylxanthines such as coca cola or Red Bull per day;
* Participation in a psychological or medical study involving the use of medication within the last 3 months;
* Previous participation in a study using the same, or similar, emotional processing tasks;
* Smoker > 10 cigarettes per day or similar levels of tobacco consumption in other forms.
* Participant received prescribed medication within 28 days prior to Visit 2 (apart from the contraceptive pill). Participants who have taken prescription medication may still be entered into the study, if, in the opinion of the Investigator, the medication received will not interfere with the study procedures or compromise safety;
* Participant received non-prescription medication, including supplements such as vitamins and herbal supplements within 48 hours prior to Visit 2 (apart from paracetamol). Participants who have taken non-prescription medication may still be entered into the study, if, in the opinion of the Investigator, the medication received will not interfere with the study procedures or compromise safety;
* Participant with a known hypersensitivity to PF-04995274, citalopram or any other serotonergic agents;
* Participant with planned medical treatment within the study period that might interfere with the study procedures;
* Participant who is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the Investigator.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Hippocampal BOLD signal during fMRI | Completed on Day 6-8
  Hippocampal and parahippocampal BOLD signal during familiar novel task - participants are presented with either previously trained (familiar) or novel images and are asked to identify whether animal or non-animal with a button press
BOLD signal during fMRI | Completed on Day 6-8
  Amygdala, anterior cingulate, prefrontal and orbitofrontal BOLD signal during emotional faces task - participants are presented with pictures of facial expressions of emotions and are asked to identify the gender of each face via button press.

SECONDARY OUTCOMES:
Auditory Verbal Learning Task (AVLT) | Completed on Day 7-9
  Accuracy of recall on the auditory verbal learning task
Emotional Memory Task | Completed on Day 7-9
  Recall and recognition of affective words displayed earlier in the testing session is tested
Facial Expression Recognition Task (FERT) | Completed on Day 7-9
  Facial expressions of basic emotions (happiness, fear, anger, disgust, sadness, surprise) are displayed on the screen and participants are asked to correctly classify them. Each emotion is presented at different intensity levels. Responses are made via a button-press and accuracy and reaction time are recorded.
Probabilistic Instrumental Learning Task (PILT) | Completed on Day 7-9
  Participants have to learn which shapes are associated with wins and losses and sensitivity to reward is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Harmer, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Murphy SE, de Cates AN, Gillespie AL, Godlewska BR, Scaife JC, Wright LC, Cowen PJ, Harmer CJ. Translating the promise of 5HT4 receptor agonists for the treatment of depression. Psychol Med. 2021 May;51(7):1111-1120. doi: 10.1017/S0033291720000604. Epub 2020 Apr 3. PMID 32241310

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT03516604/SAP_001.pdf
  • Informed Consent Form (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT03516604/ICF_000.pdf